CLINICAL TRIAL: NCT04426435
Title: Honey Based Syrup on Blood Parameters
Brief Title: Effects a Honey Based Syrup on Blood Parameters in Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Pasalar, assistant professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 22145
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; honey; blood
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Group A: patients receiving HB syrup, 10 cc three times daily
  Interventions: Drug: honey based (HB) syrup
- Placebo (Placebo Comparator): Group B: patients receiving placebo, 10 cc three times daily
  Interventions: Drug: honey based (HB) syrup

INTERVENTIONS:
Drug: honey based (HB) syrup — honey-based syrup is prepared according to the documented Persian Medicine manuscripts with some modifications. HB is a mixture of honey, rose water and saffron. Each 100g of HB consisted of 79.87 g honey, 19.97 g rose water, and 0.16 g saffron.
  All the ingredients were licensed and approved by The Islamic Republic of Iran Food and Drug Organization (I.R.I.FDO).

SUMMARY:
Study aim Determination of the effect of a honey based (HB) syrup on the blood parameters of patients with breast cancer Design Two arm parallel group randomised clinical trial, double blinded Settings and conduct Design of the study: Women patients with breast cancer referring to Shohaday-e- Tajrish Hospital of Tehran who are under chemotherapy treatment. In order to blind the investigator, medications are named as "A" for syrup of HB and B for placebo. The patients don't aware of the type of drug they are assigned to. In addition, the groups are entered into statistical analysis as "A" and "B.

The patients will revive either A or B syrup for 4 weeks. At the beginning of the trial demographic data would be gathered. Also, a blood sample would be drawn at the beginning time and after the end of intervention period (week 4).

Data would be analysed by SPSS software using T-test.

DETAILED DESCRIPTION:
Women patients with breast cancer referring to Shohaday-e- Tajrish Hospital of Tehran who are under chemotherapy treatment. In order to blind the investigator, medications are named as "A" for syrup of HB and B for placebo. The patients don't aware of the type of drug they are assigned to. In addition, the groups are entered into statistical analysis as "A" and "B.

The patients will revive either A or B syrup for 4 weeks. At the beginning of the trial demographic data would be gathered. Also, a blood sample would be drawn at the beginning time and after the end of intervention period (week 4).

Data would be analysed by SPSS software using T-test. Main outcome variables The mean of score of "Hemoglobine (Hb)", 2. The mean of score of "white blood cell count (WBC)", 3. The mean of score of "platelet count (Plt)"

Main outcome variables The mean of score of "Hemoglobine (Hb)", 2. The mean of score of "white blood cell count (WBC)", 3. The mean of score of "platelet count (Plt)"

Participants/Inclusion and exclusion criteria Inclusion criteria: women suffer from breast cancer who are; 1.Age between 18- 70 years old; 2. Hemoglobin level is at least 8g/dl; 3. Hematocrit level at least 30%; 4. normal TSH. Exclusion criteria: 1. Heart disease with unstable conditions; 2. Disabling Pulmonary Disease and History of Asthma; 3. Severe kidney disease; 4. Creatinine level greater than 2mg/dl; 5. Proteinuria; 6. The SGOT level more than 3 times of the normal threshold; 7. Bilirubin levels greater than 2mg/dl; 8. Positive history of hypersensitivity to saffron, rose water and honey; 9. severe infection; 10. Systemic disease;11. Positive history of gout or high level of uric acid; 12. An individual who uses antidepressants due to depression; 13. Simultaneous use of drugs that affect fatigue; 14. Uncontrolled pain; 15. Unwillingness to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age between 18- 70 years old Patients
* known case of breast cancer
* Hemoglobin level is at least 8 g / dl
* Hematocrit level at least 30% The level of
* TSH is normal

Exclusion Criteria:

* Patients known case of heart disease with unstable conditions
* Disabling Pulmonary Disease and History of Asthma
* Patients known case of severe kidney disease (Creatinine level is greater than 2mg / dl Proteinuria)
* The SGOT level is more than 3 times of the normal threshold
* Bilirubin levels is greater than 2mg / dl
* Positive history of hypersensitivity to saffron, Rose water and Honey
* Uncontrolled pain
* severe infection
* serious illness
* Positive history of gout or high level of uric acid
* An individual who uses antidepressants due to depression
* Simultaneous use of drugs that affect blood cells
* Unwillingness to participate in the study
* Active treatment for anemia (transfusion or Epoetin Alfa Injection)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
The change of mean score of Hemoglobin level of patients in intervention and placebo groups | The weeks of 0 and 4 after treatment
  A mean score of hemoglobin level is generally defined as 12.5 to 14.5 grams per deciliter (125-145 grams per liter) for women. Higher or lower scores mean a worse outcome.
The change of mean score of WBC count of patients in intervention and placebo groups | The weeks of 0 and 4 after treatment
  A mean score of WBC count is usually between 4,000 and 11,000 per microliter of blood for women. Higher or lower scores mean a worse outcome.
The change of mean score of Plt count of patients in intervention and placebo groups | The weeks of 0 and 4 after treatment
  A mean score of Plt count is usually ranges from 150,000 to 450,000 platelets per microliter of blood for women. Higher or lower scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Pasalar, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shohaday-e- Tajrish Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pasalar M, Choopani R, Mosaddegh M, Kamalinejad M, Mohagheghzadeh A, Fattahi MR, Ghanizadeh A, Bagheri Lankarani K. Efficacy and safety of jollab to treat functional dyspepsia: a randomized placebo-controlled clinical trial. Explore (NY). 2015 May-Jun;11(3):199-207. doi: 10.1016/j.explore.2015.02.007. Epub 2015 Feb 17. PMID 25777290
- [Result] Pasalar M, Choopani R, Mosaddegh M, Kamalinejad M, Mohagheghzadeh A, Fattahi MR, Zarshenas MM, Jafari P, Lankarani KB. Efficacy of jollab in the treatment of depression in dyspeptic patients: a randomized double-blind controlled trial. J Evid Based Complementary Altern Med. 2015 Apr;20(2):104-8. doi: 10.1177/2156587214563542. Epub 2015 Jan 13. PMID 25587004
- [Result] Emtiazy M, Oveidzadeh L, Habibi M, Molaeipour L, Talei D, Jafari Z, Parvin M, Kamalinejad M. Investigating the effectiveness of the Trigonella foenum-graecum L. (fenugreek) seeds in mild asthma: a randomized controlled trial. Allergy Asthma Clin Immunol. 2018 May 2;14:19. doi: 10.1186/s13223-018-0238-9. eCollection 2018. PMID 29743896
- [Result] Taavoni S, Fathi L, Nazem-Ekbatani N, Haghani H. The Effect of Oral Intake of Honey Syrup on the Pain Intensity of Active Phase of Parturition of nulliparous women: A Randomized clinical trial. Caspian J Intern Med. 2019 Winter;10(1):98-101. doi: 10.22088/cjim.10.1.98. PMID 30858948